CLINICAL TRIAL: NCT01205399
Title: A Single Arm, Multi-Center, Retrospective Study With Prospective Follow-Up of Complex Ventral Hernia Repair Utilizing the AlloMax Surgical Graft
Brief Title: A Retrospective Study With Prospective Follow-Up of Complex Ventral Hernia Repair Utilizing the AlloMax Surgical Graft
Acronym: AlloMax
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: DVL-HE006
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AlloMax Surgical Graft Group

SUMMARY:
This study will enroll subjects who underwent a ventral hernia repair using the AlloMax Surgical Graft at least 9 months in the past.

All subjects who underwent a ventral hernia repair using the AlloMax Surgical Graft at least 9 months in the past will be contacted and asked to take part in this clinical study. The consented subjects' medical records will be reviewed for evidence of any risk factors of hernia recurrence, procedure time, complications and any documented recurrences. The subjects will be asked to undergo a physical exam to rule out any recurrences that were not documented in the medical records.

DETAILED DESCRIPTION:
Study protocol was amended in June of 2011 to exclude further enrollment of subjects who underwent ventral hernia repair with the AlloMax Surgical Graft to bridge hernia defects.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone a ventral hernia repair using the AlloMax Surgical Graft at least 9 months in the past. (June 2011 protocol amendment further specified inclusion of subjects who have undergone a non-bridging hernia repair.)
* Have signed an informed consent form (ICF).

Exclusion Criteria:

* Underwent implantation of the AlloMax Surgical Graft for any reason other than ventral hernia repair.
* June 2011 protocol amendment added: used AlloMax Surgical Graft to bridge a defect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone a ventral hernia repair using the AlloMax Surgical Graft at least 9 months in the past.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Roth, MD, Principal Investigator — University of Kentucky
Locations (5):
- United States (5):
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Benrus Surgical Associates, Inc, City of Saint Peters, Missouri
  - Winthrop Surgical Associates, Inc., Mineola, New York
  - Surgical Associates, Inc., Tulsa, Oklahoma
  - Golla Center for Plastic Surgery, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2010 through October 2011 a total of 78 subjects were enrolled at 4 study centers in the United States. The fifth site was terminated because subject data could not be source verified.
Groups:
- AlloMax Surgical Graft Group: The study group included eligible subjects who underwent hernia repair using the AlloMax™ Surgical Graft at least 9 months prior to the start of this study.
Period: Overall Study
Arm/Group | AlloMax Surgical Graft Group
Started | 78
Completed | 78
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AlloMax Surgical Graft Group
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (11.07)
Gender [Count of Participants; unit: Participants]
  Female | 43
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 74
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 78
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] | 36.7 (9.92)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Hernia Recurrence Post Repair With an AlloMax Surgical Graft
Description: A recurrent hernia is a hernia, confirmed by the Investigator at any point after surgery, in the same location as the hernia repaired in the index procedure.
Time Frame: 9 + Months
Population: All enrolled subjects that could be verified through historical medical record review.
Measure: Number; unit: participants
Arm/Group | AlloMax Surgical Graft Group
Number analyzed (Participants) | 78
participants | 17

2. Secondary Outcome: Complications in Subjects With Hernias Repaired With an AlloMax Surgical Graft.
Description: Complications will be assessed by evaluation of the procedural and device related adverse events (AEs) documented in the subject's medical files from the time surgery was initiated until the day the subject had a postoperative visit.
Time Frame: 9+ Months
Population: All enrolled subjects that could be verified through historical medical record review.
Measure: Number; unit: complication events
Arm/Group | AlloMax Surgical Graft Group
Number analyzed (Participants) | 78
complication events | 166

3. Secondary Outcome: Procedural Time for AlloMax Surgical Graft Placement.
Description: Procedure time will be defined as beginning when the Investigator made the initial incision and ending when the skin closure was completed (skin to skin).
Time Frame: 0 Days
Population: All enrolled subjects that could be verified through historical medical record review.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AlloMax Surgical Graft Group
Number analyzed (Participants) | 78
minutes | 161.8 (58.45)

ADVERSE EVENTS:
Arm/Group | AlloMax Surgical Graft Group
Serious Adverse Events (participants affected / at risk) | 50/78
Other Adverse Events (participants affected / at risk) | 46/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlloMax Surgical Graft Group (N=78)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Impaired healing (General disorders) | 2 (2)
Abdominal abscess (Infections and infestations) | 3 (3)
Abdominal infection (Infections and infestations) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 5 (5)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3)
Clostridial infection (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 4 (4)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 12 (12)
Open wound (Injury, poisoning and procedural complications) | 3 (3)
Postoperative wound complication (Injury, poisoning and procedural complications) | 3 (3)
Seroma (Injury, poisoning and procedural complications) | 15 (16)
Suture related complication (Injury, poisoning and procedural complications) | 1 (2)
Culture wound positive (Investigations) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Caesaren section (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlloMax Surgical Graft Group (N=78)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Epidermolysis (Congenital, familial and genetic disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 16 (17)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 12 (13)
Nausea (Gastrointestinal disorders) | 12 (13)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
Pyrexia (General disorders) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 2 (2)
Body tinea (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 6 (6)
Postoperative wound infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 3 (3)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 7 (7)
Open wound (Injury, poisoning and procedural complications) | 2 (2)
Post procedural constipation (Injury, poisoning and procedural complications) | 2 (2)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 3 (3)
Seroma (Injury, poisoning and procedural complications) | 10 (10)
Blood culture positive (Investigations) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 3 (3)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1)
Scar (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was designed to use existing data. Limitations include: limited data generalizability given the retrospective, single arm, observational study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days